CLINICAL TRIAL: NCT05419076
Title: A Single Arm Phase II Study Assessing Efficacy of Stereotactic Radiosurgery (SRS) for Brain Metastasis (BM) From Small Cell Lung Cancer (SCLC)
Brief Title: A Study of Stereotactic Radiosurgery (SRS) for People With Lung Cancer That Has Spread to the Brain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-133
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer; Lung Cancer Metastatic; Brain Metastases; Brain Metastases, Adult; Small-cell Lung Cancer; Small Cell Lung Carcinoma
Keywords: Stereotactic Radiosurgery; small cell lung cancer; small cell lung carcinoma; lung cancer; lung cancer metastatic; brain metastases; 22-133; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Lung Neoplasms; Brain Neoplasms; Small Cell Lung Carcinoma | interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants with small cell lung cancer with brain metastases (Experimental): Participants may be newly diagnosed small cell lung cancer with brain metastases at initial staging, or can alternatively be patients who develop brain metastases on therapy or during surveillance of systemic disease.
  Interventions: Radiation: Stereotactic Radiosurgery; Procedure: Cerebrospinal fluid collection

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — All participants will undergo MSK standard SRS. A CT simulation will be performed per institutional standards, typically with contrast unless a contraindication exists. A contrast-enhanced MRI with 1mm slices will be fused to the CT simulation scan for the purposes of SRS planning. The SRS GTV will be considered the visible tumor on MRI and CT contrast enhanced studies. An expansion of 1-2mm will be used to create the PTV. Radiation dose may be between 16Gy and 30Gy in 1 to 5 fractions, per the discretion of the treating radiation oncologist. Participants with multiple lesions may receive different doses to each lesion per the discretion of the treating radiation oncologist. Concurrent treatment to other body sites is permitted.
  Other Names: SRS
Procedure: Cerebrospinal fluid collection — All participants will undergo lumbar puncture for CSF collection at study enrollment.. Lumbar punctures will be performed by clinical staff in neurology or neuroradiology, per the discretion of the treating radiation oncologist, as dictated by scheduling limitations and expected clinical difficulty in obtaining a sample (e.g. requiring fluoroscopic guidance), with input from the PI, neurology, and/or neuroradiology as necessary. Participants will be encouraged to undergo repeat lumbar puncture for CSF collection at 3 months (+/- 4 weeks), and at the time of CNS disease progression, though these latter timepoints are not required. CSF cytology will be evaluated.
  Other Names: CSF

SUMMARY:
The purpose of the study is to see if stereotactic radiosurgery/SRS is an effective treatment for people with a new diagnosis of brain metastases from small cell lung cancer/SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of small cell lung cancer
* Radiographic diagnosis of up to 20 brain metastases on contrast-enhanced MRI
* Age 18 and above
* Performance status KPS 60-100/ECOG 0-2
* Female patients must be of non-reproductive potential or have a negative serum pregnancy test at the time of enrollment
* The patient or legally authorized representative is able to provide informed consent

Exclusion Criteria:

* Unable to undergo contrast-enhanced MRI brain
* Leptomeningeal disease confirmed on lumbar puncture, MRI brain, or MRI spine
* Pregnant or lactating women
* Prior brain-directed radiotherapy
* Uncontrolled systemic disease without reasonable systemic therapy options felt likely to result in death as observed on CT or PET/CT imaging, no more than 3 months before study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 6 months
  The primary endpoint of this study is the rate of overall survival at 6 months, with time measured from the start of SRS treatment. Participants will be censored at the date of last follow up or the last date the participant was known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Luke Pike, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau, Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org